CLINICAL TRIAL: NCT04784143
Title: A Phase 2, Open-Label, Randomized Comparative Effectiveness Study for MDMA-Assisted Psychotherapy in U.S. Veterans With Chronic PTSD
Brief Title: Study Comparing Two Versus Three Active MDMA-assisted Sessions in U.S. Military Veterans With Chronic PTSD
Acronym: MPVA6
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early by the sponsor due to administrative, non-safety related reasons.
Sponsor: Lykos Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPVA6
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Results first posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2025-06

CONDITIONS: PTSD
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Psychotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Two sessions of MDMA-assisted therapy (Active Comparator): Two experimental sessions of MDMA-assisted therapy
  Interventions: Drug: Midomafetamine; Behavioral: Psychotherapy
- Three sessions of MDMA-assisted therapy (Active Comparator): Three experimental sessions of MDMA-assisted therapy
  Interventions: Drug: Midomafetamine; Behavioral: Psychotherapy

INTERVENTIONS:
Drug: Midomafetamine — 120 mg midomafetamine HCl followed by a supplemental dose of 60 mg
  Other Names: 3,4-methylenedioxymethamphetamine; MDMA; midomafetamine HCl
Behavioral: Psychotherapy — Manualized psychotherapy performed by therapist team

SUMMARY:
The goal of this clinical trial is to learn if MDMA-assisted therapy is effective in U.S. military veterans with at least moderate chronic PTSD. The main question it aims to answer is: Are two versus three MDMA-assisted therapy sessions in an outpatient treatment clinic more effective?

Researchers will compare two MDMA-assisted therapy sessions to three MDMA-assisted therapy sessions.

Participants will undergo three non-drug preparatory sessions prior to their first MDMA-assisted therapy session. Each MDMA-assisted therapy session will be followed by three non-drug integrative therapy sessions.

DETAILED DESCRIPTION:
This open-label, randomized study will assess the comparative effectiveness of two versus three active MDMA-assisted therapy sessions in U.S. military veterans with at least moderate chronic PTSD treated in an outpatient VA treatment clinic. The study will be conducted in up to 60 participants. Prior to the randomized portion of the study, each therapist pair team will treat one participant under the 3-session model, and one participant under the 2-session model. In total, 8 participants will be treated under this proof of principle therapist training lead-in. A 120 mg dose of MDMA, followed by a supplemental dose (60 mg) unless contraindicated, is administered during the treatment period with manualized psychotherapy in 2 or 3 open-label monthly Experimental Sessions. This ~ 8-12-week Treatment Period includes three Preparatory Sessions prior to the first MDMA-assisted session. During the treatment period, each Experimental Session is followed by three Integrative Sessions of non-drug therapy. The Primary Outcome measure, the Clinician-Administered PTSD Scale for DSM-5 (CAPS-5), is assessed by a centralized, blinded Independent Rater (IR) pool at post-treatment for each group.

ELIGIBILITY:
Inclusion Criteria:

* U.S. military veteran
* Are at least 18 years old.
* Are fluent in speaking and reading the predominantly used or recognized language of the study site.
* Are able to swallow pills.
* Agree to have study visits recorded, including Experimental Sessions, Independent Rater assessments, and non-drug psychotherapy sessions.
* Must provide a contact (relative, spouse, close friend or other caregiver) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
* Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
* If of childbearing potential, must have a negative pregnancy test at study entry and prior to each Experimental Session, and must agree to use adequate birth control through 10 days after the last Experimental Session.
* Must not participate in any other interventional clinical trials during the duration of the study.
* Must be willing to remain overnight at the study site after each Experimental Session and be driven home after, and commit to medication dosing, therapy, and study procedures.
* At baseline, have moderate PTSD diagnosis.

Exclusion Criteria:

* Are not able to give adequate informed consent.
* Have uncontrolled hypertension.
* Have a marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 milliseconds [ms] corrected by Bazett's formula).
* Have a history of additional risk factors for Torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome).
* Have evidence or history of significant medical disorders.
* Have symptomatic liver disease.
* Have history of hyponatremia or hyperthermia.
* Weigh less than 48 kilograms (kg).
* Are pregnant or nursing, or are of childbearing potential and are not practicing an effective means of birth control.
* Have used Ecstasy (material represented as containing MDMA) more than 10 times within the last 10 years or at least once within 6 months of the first Experimental Session; or have previously participated in a MAPS-sponsored MDMA clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-11-08 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Yehuda, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- James J. Peters VA Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Two Sessions of MDMA-assisted Therapy | Three Sessions of MDMA-assisted Therapy
Started | 13 | 10
Completed | 12 | 8
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Two Sessions of MDMA-assisted Therapy | Three Sessions of MDMA-assisted Therapy | Total
Number analyzed (Participants) | 13 | 10 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (6.23) | 38.3 (5.06) | 40.2 (5.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 12 | 10 | 22
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 10 | 6 | 16
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 9 | 8 | 17
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 13 | 10 | 23
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Score [Mean (Standard Deviation); unit: score on a scale] — The CAPS-5 is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values indicating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.
  score on a scale | 37.1 (6.38) | 43.8 (7.71) | 40.0 (7.63)

OUTCOME MEASURES:

1. Primary Outcome: Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score From Baseline to Primary Outcome
Description: The Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values indicating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.
Time Frame: 2 Session Group: ~12 weeks from baseline to primary outcome; 3 Session Group: ~16 weeks from baseline to primary outcome
Population: One participant in the 3 session group did not complete the primary outcome assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Two Sessions of MDMA-assisted Therapy | Three Sessions of MDMA-assisted Therapy
Number analyzed (Participants) | 13 | 9
score on a scale | -20.5 (9.38) | -18.0 (13.92)

2. Primary Outcome: Change in Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) Total Severity Score From Baseline to Secondary Outcome Timepoint in the 2 Session Group
Description: as for outcome 1
Time Frame: ~16 weeks from baseline to secondary outcome (note: secondary outcome timepoint assessed in 2 session group to evaluate the primary outcome measure in a follow up period equivalent to that of the 3 session group in the primary analysis.)
Population: One participant in the 2 session group did not complete the CAPS-5 at the secondary outcome timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Two Sessions of MDMA-assisted Therapy
Number analyzed (Participants) | 12
score on a scale | -24.9 (8.73)

3. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score From Baseline to Primary Outcome
Description: The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities, with each item scored on a ten-point Likert scale from 0 ('not at all impaired') to 10 ('very severely impaired'). SDS scoring was adapted for the purposes of this study to limit missing item-level data through averaging the three domain scores to produce a total score, as well as imputation of work-related impairment score in the case of participants who did not work during the reporting period based on the reason for not working. The SDS total score and each of the domain sub-scores range from 0 to 10, with higher scores indicating greater functional impairment.
Time Frame: as for outcome 1
Population: One participant in the 3 session group did not complete the secondary outcome assessment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Two Sessions of MDMA-assisted Therapy | Three Sessions of MDMA-assisted Therapy
Number analyzed (Participants) | 13 | 9
score on a scale | -2.9 (2.30) | -1.6 (3.49)

4. Secondary Outcome: Change in Sheehan Disability Scale (SDS) Total Score From Baseline to Secondary Outcome Timepoint in the 2 Session Group
Description: Sheehan Disability Scale (SDS) total score, a measure of clinician-rated functional impairment. The items indicate degree of impairment in the domains of work/school, social life, and home life, with response options based on an eleven-point scale (0=not at all to 10=extremely), and five verbal tags (not at all, mildly, moderately, markedly, extremely).
Time Frame: as for outcome 2
Population: One participant in the 2 session group did not complete the SDS at the secondary outcome timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Two Sessions of MDMA-assisted Therapy
Number analyzed (Participants) | 12
score on a scale | -4.1 (2.39)

ADVERSE EVENTS:
Time Frame: During the Treatment Period from the first Experimental Session to the Termination visit (2-session group: approximately 13 weeks, 3-session group: approximately 16 weeks)
Arm/Group | Two Sessions of MDMA-assisted Therapy | Three Sessions of MDMA-assisted Therapy
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/10
Other Adverse Events (participants affected / at risk) | 13/13 | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Two Sessions of MDMA-assisted Therapy (N=13) | Three Sessions of MDMA-assisted Therapy (N=10)
Insomnia (Psychiatric disorders) | 10 | 5
Bruxism (Psychiatric disorders) | 7 | 4
Depressed mood (Product Issues) | 2 | 3
Agitation (Psychiatric disorders) | 2 | 1
Anger (Psychiatric disorders) | 2 | 1
Fear (Psychiatric disorders) | 2 | 1
Irritability (Psychiatric disorders) | 2 | 1
Nightmare (Psychiatric disorders) | 1 | 2
Restlessness (Psychiatric disorders) | 3 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 2
Feeling guilty (Psychiatric disorders) | 0 | 2
Illusion (Psychiatric disorders) | 1 | 1
Affect lability (Psychiatric disorders) | 1 | 0
Attention deficit hyperactivity disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Derealisation (Psychiatric disorders) | 0 | 1
Dissociation (Psychiatric disorders) | 0 | 1
Dysphoria (Psychiatric disorders) | 0 | 1
Emotional disorder (Psychiatric disorders) | 1 | 0
Feeling of despair (Psychiatric disorders) | 0 | 1
Flashback (Psychiatric disorders) | 1 | 0
Flight of ideas (Psychiatric disorders) | 0 | 1
Intrusive thoughts (Psychiatric disorders) | 1 | 0
Loss of libido (Psychiatric disorders) | 0 | 1
Panic attack (Psychiatric disorders) | 0 | 1
Panic reaction (Psychiatric disorders) | 0 | 1
Poor quality sleep (Psychiatric disorders) | 0 | 1
Suicidal behaviour (Psychiatric disorders) | 0 | 1
Tic (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 3 | 3
Headache (Nervous system disorders) | 5 | 8
Nystagmus (Nervous system disorders) | 3 | 3
Dizziness (Nervous system disorders) | 1 | 3
Disturbance in attention (Nervous system disorders) | 0 | 3
Paraesthesia (Nervous system disorders) | 1 | 2
Hypoaesthesia (Nervous system disorders) | 1 | 1
Tremor (Nervous system disorders) | 1 | 1
Head discomfort (Nervous system disorders) | 1 | 0
Lethargy (Nervous system disorders) | 0 | 1
Parosmia (Nervous system disorders) | 0 | 1
Presyncope (Nervous system disorders) | 1 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 2 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Feeling of relaxation (General disorders) | 2 | 5
Feeling cold (General disorders) | 3 | 3
Feeling hot (General disorders) | 1 | 5
Therapeutic response unexpected (General disorders) | 3 | 2
Fatigue (General disorders) | 1 | 3
Chest discomfort (General disorders) | 1 | 1
Thirst (General disorders) | 2 | 0
Chills (General disorders) | 0 | 1
Feeling abnormal (General disorders) | 0 | 1
Feeling drunk (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 3 | 5
Nausea (Gastrointestinal disorders) | 3 | 5
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Anal paraesthesia (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Lip swelling (Gastrointestinal disorders) | 0 | 1
Proctalgia (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Mydriasis (Eye disorders) | 3 | 5
Photophobia (Eye disorders) | 3 | 3
Visual impairment (Eye disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Blood pressure increased (Investigations) | 4 | 4
Decreased appetite (Metabolism and nutrition disorders) | 5 | 1
Alcohol intolerance (Metabolism and nutrition disorders) | 0 | 1
Food craving (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 3
Dysuria (Renal and urinary disorders) | 0 | 1
Urinary hesitation (Renal and urinary disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperventilation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Yawning (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 1
Cold sweat (Skin and subcutaneous tissue disorders) | 2 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Ear discomfort (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Genital pain (Reproductive system and breast disorders) | 0 | 1
Substance use (Social circumstances) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-08-04): https://cdn.clinicaltrials.gov/large-docs/43/NCT04784143/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-18): https://cdn.clinicaltrials.gov/large-docs/43/NCT04784143/SAP_001.pdf